CLINICAL TRIAL: NCT04635046
Title: Effects on Patient Satisfaction and Gait After Loss of Peroneus Longus Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Anna Sprinchorn (Other)
Responsible Party: Sponsor-Investigator, Anna Sprinchorn, Principal Investigator, Uppsala University
Organization: Uppsala University (Other)
Other Study IDs: 2015/428
Record Dates: First submitted 2020-09-18; First posted 2020-11-18 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Patient Satisfaction; Gait, Rigid
Keywords: Cavovarus foot; Gait analysis; Tendon transfer
MeSH Terms: conditions — Patient Satisfaction; Gait Disorders, Neurologic | interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with tears to their peroneal tendons: Patients with pain over their peroneal tendons clinically, with a verified injury to either of the two tendons on MRI, where we might expect a tendon transfer of the peroneus longus, or extirpation of the peroneus longus, during surgery.
  Interventions: Procedure: Transfer or extirpation of the peroneus longs tendon

INTERVENTIONS:
Procedure: Transfer or extirpation of the peroneus longs tendon — Tendon transfer or extirpation of peroneus longus or brevis tendon, ligamental reconstruction +/- calcaneal osteotomy

SUMMARY:
At the foot and ankle group at the Department of Orthopaedics, Uppsala University Hospital, the routine is to perform a tendon transfer of peroneus longus to brevis in case of a ruptured peroneus brevis tendon in the ankle. The reports of patient outcome from this surgery varies in different studies. The aim of the current study is to analyse how well the patients think their general health has improved after the surgery, and how they perceive that the foot function has changed after the surgery. In an objective way the changes in gait after surgery will be measured with gait analysis.

DETAILED DESCRIPTION:
The patients are asked to fill in Short Form 36 (SF 36) and Foot and Ankle Outcome Score (FAOS) before surgery, six months and one year after surgery. At each visit a clinical examination is done by a foot and ankle surgeon, according to a protocol. At the same visit a gait analysis is performed with force plates, registration of speed and gait length and 3D recording. The surgery itself is performed according to the clinic's usual protocol and standardised, so all patients are treated in the same way. The physiotherapy is also done according to a protocol. The surgeon is not involved in the follow- up, this is done by another surgeon, and the gait analysis is done by a physiotherapist.

The patients are chosen from two groups: primary tear of the peroneus brevis tendon, requiring a longus to brevis transfer, and primary tear of the peroneus longus tendon, requiring removal of the tendon.

The first group has a sub-group: patients who are in need of a calcaneal osteotomy because of a severe varus hindfoot. The reason the study group is so heterogenous is that peroneus longus and brevis tears are very rare, and 10 patients are referred to the Orthoaedic deparment each year, that need this type of surgery. The sample size has been calculated to 30 patients (based on changes in force measurements during gate), but more patients need to be involved in the study in order to have 30 patients at one year follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Tears of the peroneus longus and/or peroneus brevis tendon, verified on MRI.
2. Eligible for surgery of peroneal tendon tears

Exclusion Criteria:

1. Other injuries in the affected foot that might affect the gait.
2. Previous surgery in the affected foot that might affect the gait.
3. Neurological conditions in the lower extremities that might affect the gait.
4. Patient can not understand the questionnaires or can not understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are referred to the Foot and Ankle Clinic at Uppsala University Hospital with a tear to the peroneus brevis or longus tendon where we plan for surgery, and who are willing to participate in the study after information about the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life one year after foot surgery including a peroneus longus transfer | Before surgery to 12 months after surgery
  Patients quality of life is measured with the self-administered Short Form 36 ( SF 36 ) (range 0-100 points, 100 points best health) before surgery, at 6 months and 12 months after surgery.
Changes in foot function one year after surgery including a peroneus longus transfer | Before surgery to 12 months after surgery
  Changes in foot function after surgery is measured using a patient reported outcome measure: Foot and Ankle Outcome Score (FAOS) (range 0-100 points, 100 points being a totally healthy foot). The patient fill in the score before surgery, at 6 months and 12 months after surgery.

SECONDARY OUTCOMES:
Weakness in push-off during gait | One year after surgery
  After removal of the peroneus longus tendon one might observe a weakness in the plantar flexion of the first metatarsal bone, leading to a weakness in push off during gait. This will be measured on the RSscan pressure mat (from RSscan International), recording the pressure at push-off in Newtons/ m2. The patient will be walking both bare foot and with shoes. Measurements are done before surgery, at 6 months and 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Michaelsson, PhD, Study Chair — Professor
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04635046/Prot_SAP_000.pdf